CLINICAL TRIAL: NCT00587158
Title: Oral Paricalcitol in Kidney Transplant Recipients Receiving a Corticosteroid-free Immunosuppressive Regimen
Brief Title: Oral Paricalcitol in Kidney Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Hatem Amer, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 256-06
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2013-05-08 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Transplant; Failure, Kidney; Renal Disease, End Stage; Hyperparathyroidism, Secondary
Keywords: Paricalcitol; Parathyroid Hormone; Bone Alkaline Phosphatase; Chronic Kidney Disease; Glomerular Filtration Rate; Vitamin D Receptor; Interstitial Fibrosis and Tubular Atrophy; Zemplar®
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic; Pulmonary Fibrosis | interventions — paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immunosuppression without paricalcitol (control) (Other): Subjects will receive the standard immunosuppressive therapies consisting of induction therapy with Alemtuzumab (Campath®) and Methylprednisolone (Solumedrol®), then maintained with corticosteroid avoidance using Mycophenolate Mofetil (Cellcept®) and Tacrolimus (Prograf®).
  Interventions: Other: Corticosteroid Avoidance Immune Suppression Protocol
- Immunosuppression with paricalcitol (Active Comparator): Subjects will receive the standard immunosuppressive therapy consisting of induction therapy with Alemtuzumab (Campath®) and Methylprednisolone (Solumedrol®), then maintained with corticosteroid avoidance using Mycophenolate Mofetil (Cellcept®) and Tacrolimus (Prograf®). In addition, subjects will receive the study medication paricalcitol (Zemplar®).
  Interventions: Drug: Paricalcitol; Other: Corticosteroid Avoidance Immune Suppression Protocol

INTERVENTIONS:
Drug: Paricalcitol — Zemplar® - this medicine, which is the medicine being studied, will be given as a capsule containing 1 microgram of Zemplar® once daily beginning the day after the transplant. It will be continued at the same dose for the first two weeks then, depending on the results of blood and urine testing, will be increased to 2 micrograms daily. The dose will remain at 2 micrograms daily until the end of the study unless there is a medical reason to reduce or stop it or unless the study is stopped early.
  Other Names: Brand name is Zemplar®
  Arms: Immunosuppression with paricalcitol
Other: Corticosteroid Avoidance Immune Suppression Protocol — Induction with Alemtuzumab and maintenance with Tacrolimus and Mycophenolate Mofetil. With standard antimicrobial prophylaxis and calcium supplementation.
  Other Names: Standard Immune Suppression

SUMMARY:
This study is being done to find out whether patients who receive a kidney transplant can benefit from taking the medication paricalcitol (trade name Zemplar®) as compared to kidney transplant recipients not taking this medication. The main possible benefits being studied are:

* Lower risk for overactive parathyroid glands after kidney transplantation.
* Lower risk of low bone density in the spine and hip after kidney transplantation. By dividing patients in the study into a group receiving Zemplar® and a group not receiving Zemplar®, it will be possible to understand the good and bad effects of Zemplar® during the first year after a kidney transplant.

DETAILED DESCRIPTION:
The most significant challenge in kidney transplantation at present is that of reducing the risk of long-term complications. This includes hyperparathyroidism, a common post kidney transplant complication that contributes to loss of bone density and fracture risk and necessitates surgical intervention in approximately 5% of kidney transplant patients.

In order to take part in the study you will already have been accepted for kidney transplantation from a living donor or from a deceased donor at Mayo Clinic in Rochester, Minnesota. After you have agreed to take part in the study you will be put in one of two groups by chance (as in the flip of a coin):

Group 1 (Standard Treatment or "Control"): Patients in this group will receive a combination of four anti-rejection medications that have been used at Mayo Clinic Rochester for many kidney transplant patients and does not include any research study medicines. These medications will include:

1. Alemtuzumab (Campath®) - this medicine will be given intravenously (IV) on the day of the transplant during surgery.
2. Methylprednisolone (Solumedrol®) - this medicine, which is part of a family of medicines often referred to as corticosteroids, will be given intravenously on the day of the transplant during surgery. This will be the only planned dose of corticosteroid medicine you will receive although this medicine and a tablet form called Prednisone may be given at a later time if you have an episode of transplant rejection.
3. Mycophenolate Mofetil (Cellcept®) - this medicine will be given by mouth twice daily beginning the evening before the transplant (for living donor transplants) or the day of the transplant (for deceased donor transplants). It will be continued for as long as you have your transplant unless there is a medical reason to stop it.
4. Tacrolimus (Prograf®) - this medicine will be given by mouth once daily beginning on the fourth day after the transplant. It will continue for as long as you have your transplant unless there is a medical reason to stop it. The dose will be adjusted based on a blood test that will be done between twice a week and once a month for as long as you take the medicine.

Group 2 (Zemplar® + Standard Treatment): Patients in this group will receive the same combination of anti-rejection medications as the patients in Group 1 (a-d above) plus Zemplar®, which is the medicine being studied, will also be started on the day of the transplant. Zemplar® will be given as a capsule containing 1 microgram of Zemplar® once daily beginning the day after the transplant. It will be continued at the same dose for the first two weeks then, depending on the results of blood and urine testing, will be increased to 2 micrograms daily. The dose will remain at 2 micrograms daily until the end of the study unless there is a medical reason to reduce or stop it or unless the study is stopped early.

Both groups of patients will be treated by the same team of doctors, nurses and nurse coordinators that care for all kidney transplant patients at Mayo Clinic. The procedures and treatments for your transplant will be the same as those recommended at Mayo Clinic for all patients receiving a kidney transplant. These include the surgical operation to carry out the transplant; the need to take anti-rejection medicines by mouth for the rest of your life; the need to have blood and urine testing at regular intervals for the rest of your life to monitor the progress of your transplant; and the recommendation to have a biopsy of your transplant carried out on three occasion during the first two years after the transplant surgery. These procedures and their potential complications will be described to you in detail by your transplant physician, transplant surgeon, and transplant coordinator. The study will not require extra hospital or outpatient visits compared to the usual care for all kidney transplant patients at Mayo Clinic Rochester.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older.
* First or second deceased donor or living donor renal transplant.
* Normocalcemia or hypocalcemia.
* Willing to give informed consent

Exclusion Criteria:

* Third or subsequent renal transplant.
* Incompatible blood type or positive cross-match donor.
* Multiple organ transplant recipients.
* Diabetic with plans for future pancreas or islet transplant.
* Evidence of donor-specific sensitization (positive T-cell and/or B-cell flow cytometric cross-match).
* Documented hypercalcemia (total serum calcium 10.5 mg/dl on two separate occasions) prior to transplantation.
* Serum 25(OH)vitamin D concentration ≤ 10 ng/ml

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Amer, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients to undergo kidney transplantation at Mayo Clinic facilities in Rochester, Minnesota and in Scottsdale, Arizona and scheduled to receive corticosteroid avoidance anti-rejection therapy were screened for enrollment into the study.
Pre-assignment Details: 112 patients were approached for enrollment. Of those, 4 patient's treating physicians did not think corticosteroid free immunosuppression was appropriate, 3 had their transplants cancelled, 3 were found to be vitamin D deficient, 1 withdrew consent prior to randomization & 1 had a positive final crossmatch and hence were excluded from the study.
Groups:
- Immunosuppression With Paricalcitol: Subjects will receive the standard immunosuppressive therapy consisting of induction therapy with Alemtuzumab (Campath®) and Methylprednisolone (Solumedrol®), then maintained with corticosteroid avoidance using Mycophenolate Mofetil (Cellcept®) and Tacrolimus (Prograf®). In addition, subjects in this group will receive the study medication paricalcitol (Zemplar®).
Period: Overall Study
Arm/Group | Immunosuppression Without Paricalcitol (Control) | Immunosuppression With Paricalcitol
Started | 49 | 51
Continued in Study | 45 | 46
Completed | 44 | 43
Not Completed | 5 | 8
Not completed — Did not want to do 24 hr urine collect. | 4 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Death | 0 | 1
Not completed — Subject did not want to take study med | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Immunosuppression Without Paricalcitol (Control): Subjects will receive the standard immunosuppressive therapies of Alemtuzumab (Campath®), Methylprednisolone (Solumedrol®), Mycophenolate Mofetil (Cellcept®) and Tacrolimus (Prograf®).
- Immunosuppression With Paricalcitol: Subjects will receive the standard immunosuppressive medications; Alemtuzumab (Campath®), Methylprednisolone (Solumedrol®),Mycophenolate Mofetil (Cellcept®) and Tacrolimus (Prograf®), and in addition will receive the study medication paricalcitol (Zemplar®).
- Total: Total of all reporting groups
Arm/Group | Immunosuppression Without Paricalcitol (Control) | Immunosuppression With Paricalcitol | Total
Number analyzed (Participants) | 49 | 51 | 100
Age Continuous [Mean (Standard Deviation); unit: years] | 47.7 (10.0) | 48.5 (10.3) | 48.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 33 | 33 | 66
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 0 | 3
  White | 42 | 49 | 91
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
  Hispanic | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 49 | 51 | 100
Diabetes [Number; unit: participants] — Not all subjects were diabetic, so the total number of subjects within each arm will not match the number of subjects with diabetes within each arm.
  participants | 12 | 10 | 22
First transplant [Number; unit: participants] — Because this was not the first transplant for some subjects, the number of subjects having their first transplant will not match the total number of subjects in each arm.
  participants | 47 | 50 | 97
Cause of End-Stage Renal Disease [Number; unit: participants]
  Adult Polycystic Kidney Disease | 14 | 16 | 30
  Diabetic | 10 | 8 | 18
  Glomerulonephritis | 17 | 16 | 33
  Hypertension | 1 | 3 | 4
  Other | 7 | 8 | 15
Living kidney donor [Number; unit: participants] — Because some of the donor kidneys were from cadaver donors, the number of subjects receiving a kidney from living donors will not match the total number of subjects in each arm.
  participants | 48 | 48 | 96
Degree of interstitial fibrosis [Number; unit: Participants] — Interstitial fibrosis refers to degree of scarring or fibrous tissue formed in the kidney. Renal pathologists reviewed biopsies of the subject's kidney grafts for fibrosis, with results expressed according to the Banff schema. The degree of fibrosis was reported using Banff scores (ci) as "mild" (ci greater than 0 and less than 2) or "moderate to severe" (ci greater than or equal to 2). Because not all subjects had interstitial fibrosis in their kidneys, the number with fibrosis will differ from the overall number of subjects in each treatment group.
  Participants
    Mild fibrosis at baseline | 2 | 3 | 5
    Moderate to severe fibrosis at baseline | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Hyperparathyroidism at One Year
Description: Parathyroid hormone (PTH) is a measure of how well the parathyroid gland is working and is measured by a blood test. Hyperparathyroidism (increased PTH) is defined as PTH blood value greater than 65 picograms/milliliter in the absence of hypocalcemia (low calcium) or if the subject had a parathyroidectomy (surgical removal of parathyroid glands) during the first year post-transplant.
Time Frame: 1 year post kidney transplant
Population: Analysis was performed by the intention-to-treat principle, comprised of all subjects enrolled, who will have taken at least one dose of study medication and have both screening and any post-screening efficacy data recorded. The last observation was carried forward for missing values.
Measure: Number; unit: Participants
Arm/Group | Immunosuppression Without Paricalcitol (Control) | Immunosuppression With Paricalcitol
Number analyzed (Participants) | 49 | 51
Participants | 31 | 15
Statistical Analysis 1: Comparison: Immunosuppression Without Paricalcitol (Control) vs Immunosuppression With Paricalcitol; Test type: Superiority or Other; p = 0.0005, Fisher Exact

2. Secondary Outcome: Number of Subjects With Osteopenia/Osteoporosis of the Hip at One Year
Description: Osteopenia/Osteoporosis are conditions where bone mineral density is lower than normal, reported by T-scores, measurements of the hip made using an Dual Energy X-ray Absorptiometry (DEXA) scan. The T-score is measured and compared to a normal healthy adult. A normal bone density results in a T-score between +1.0 and -1.0. A T-score of less than or equal to -1.5 was used for this study to define the presence of osteopenia/osteoporosis. Each participant will be categorized as having or not having osteopenia/osteoporosis of the hip at the end of the first post-transplant year based on bone mineral density results.
Time Frame: 1 year post kidney transplant
Population: Per-protocol analysis. Data were not available for 2 control subjects and 2 treatment subjects, as these subjects did not have the DEXA scan of the hip done at one year. [Control n=42/ Treatment=41]
Measure: Number; unit: Participants
Arm/Group | Immunosuppression Without Paricalcitol (Control) | Immunosuppression With Paricalcitol
Number analyzed (Participants) | 42 | 41
Participants | 9 | 12
Statistical Analysis 1: Comparison: Immunosuppression Without Paricalcitol (Control) vs Immunosuppression With Paricalcitol; Test type: Superiority or Other; p = 0.4571, Fisher Exact

3. Secondary Outcome: Number of Subjects With Osteopenia/Osteoporosis of the Lumbar Spine at One Year
Description: Osteopenia/Osteoporosis are conditions where bone mineral density is lower than normal, reported by T-scores, measurements of the lower spine made using an Dual Energy X-ray Absorptiometry (DEXA) scan. The T-score is measured and compared to a normal healthy adult. A normal bone density results in a T-score between +1.0 and -1.0. A T-score of less than or equal to -1.5 was used for this study to define the presence of osteopenia/osteoporosis. Each participant will be categorized as having or not having osteopenia/osteoporosis of the lumbar spine at the end of the first post-transplant year based on bone mineral density results.
Time Frame: 1 year post kidney transplant
Population: Per-protocol analysis; Data were not available for 1 subject from each arm because these subjects did not have the one year DEXA scan of the spine. [Control n = 43/Treatment n = 42].
Measure: Number; unit: Participants
Arm/Group | Immunosuppression Without Paricalcitol (Control) | Immunosuppression With Paricalcitol
Number analyzed (Participants) | 43 | 42
Participants | 9 | 14
Statistical Analysis 1: Comparison: Immunosuppression Without Paricalcitol (Control) vs Immunosuppression With Paricalcitol; Test type: Superiority or Other; p = 0.2290, Fisher Exact

4. Secondary Outcome: Serum Parathyroid Hormone (PTH) Level Over Time
Description: Parathyroid hormone (PTH) is a hormone synthesized in the body's parathyroid glands that controls bone health. PTH controls calcium and phosphorus levels in the body. It is measured in the serum and reported in picograms per milliliter (pg/mL).
Time Frame: Baseline, 3 weeks, 3 months, 1 year post kidney transplant
Population: Per-protocol analysis; the number of samples obtained at each time point varied because not all subjects were able to undergo laboratory testing at the specified timepoints. The number of subjects samples per treatment group were as follows [Timepoint: Control(n)/Treatment(n)]:
  Baseline: 43/41, Day 21: 44/41, Day 90: 44/43, Day 365: 44/43
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Immunosuppression Without Paricalcitol (Control) | Immunosuppression With Paricalcitol
Number analyzed (Participants) | 44 | 43
pg/mL
  Baseline PTH level | 236 [50.12 to 1048.00] | 198 [55.00 to 1266.00]
  21 day PTH level | 69 [26.00 to 414.00] | 50 [11.00 to 222.00]
  3 month PTH level | 70 [34.74 to 273.00] | 42 [15.00 to 213.00]
  1 year PTH level | 85 [18.00 to 460.00] | 42 [12.00 to 266.00]
Statistical Analysis 1: Comparison: Immunosuppression Without Paricalcitol (Control) vs Immunosuppression With Paricalcitol; The median PTH level at baseline was compared between the two treatment groups; Test type: Superiority or Other; p = 0.17, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Immunosuppression Without Paricalcitol (Control) vs Immunosuppression With Paricalcitol; The median PTH level at 21 days was compared between the two treatment groups; Test type: Superiority or Other; p = 0.005, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Immunosuppression Without Paricalcitol (Control) vs Immunosuppression With Paricalcitol; The median PTH level at 90 days was compared between the two treatment groups; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Immunosuppression Without Paricalcitol (Control) vs Immunosuppression With Paricalcitol; The median PTH level at one year was compared between the two treatment groups; Test type: Superiority or Other; p = 0.0004, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Serum Bone Alkaline Phosphatase (BAP) Level Over Time
Description: BAP is a marker of bone turn-over, is measured in the serum and reported in micrograms per liter (mcg/L).
Time Frame: Baseline, 21 days, 90 days and 1 year post kidney transplant
Population: Per-protocol analysis; the number of samples obtained at each time point varied because not all subjects were able to undergo laboratory testing at the specified study visits. The number of subjects samples per treatment group were as follows [Timepoint: Control(n)/Treatment(n)]:
  Baseline: 43/41, Day 21: 34/38, Day 90: 36/36, Day 365: 43/41
Measure: Median (Full Range); unit: mcg/L
Arm/Group | Immunosuppression Without Paricalcitol (Control) | Immunosuppression With Paricalcitol
Number analyzed (Participants) | 44 | 43
mcg/L
  Baseline BAP | 14 [6.4 to 34.00] | 13 [4.9 to 50.0]
  Day 21 BAP | 16.5 [6.4 to 81.0] | 17 [3.8 to 74.0]
  Day 90 BAP | 21 [5.8 to 66.0] | 12 [3.5 to 116.0]
  Day 365 BAP | 14 [2.0 to 54.0] | 11 [4.4 to 100.0]
Statistical Analysis 1: Comparison: Immunosuppression Without Paricalcitol (Control) vs Immunosuppression With Paricalcitol; The median BAP level at baseline was compared between the two treatment groups; Test type: Superiority or Other; p = 0.833, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Immunosuppression Without Paricalcitol (Control) vs Immunosuppression With Paricalcitol; The median BAP level at 21 days was compared between the two treatment groups; Test type: Superiority or Other; p = 0.553, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Immunosuppression Without Paricalcitol (Control) vs Immunosuppression With Paricalcitol; The median BAP level at 90 days was compared between the two treatment groups; Test type: Superiority or Other; p = 0.035, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Immunosuppression Without Paricalcitol (Control) vs Immunosuppression With Paricalcitol; The median BAP level at one year was compared between the two treatment groups; Test type: Superiority or Other; p = 0.171, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Lumbar Spine Bone Mineral Density (BMD)
Description: BMD was measured using a Dual Energy X-ray Absorptiometry (DEXA) scan and reported by T-scores, measurements of the lower spine made using the scan. The T-score reflects how your bone density measurement compares to normal healthy adults. A normal bone density results in a T-score between +1.0 and -1.0. A T-score of less than or equal to -1.5 was used for this study to define the presence of osteopenia/osteoporosis. Osteopenia is a condition of decreased bone mass or density but not thin enough to be diagnosed as osteoporosis. Osteoporosis is a condition where bone mass/density has diminished to a level causing higher risk of fracture. The average change in T-score from baseline to one year is reported.
Time Frame: Baseline, 1 year post kidney transplant
Population: Per-protocol analysis; Not all subjects were able to undergo the DEXA scan of the spine at baseline and one-year [Control n = 42/Treatment n = 41].
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Immunosuppression Without Paricalcitol (Control) | Immunosuppression With Paricalcitol
Number analyzed (Participants) | 42 | 41
T-score | 0.35 (0.45) | 0.35 (0.58)
Statistical Analysis 1: Comparison: Immunosuppression Without Paricalcitol (Control) vs Immunosuppression With Paricalcitol; Test type: Superiority or Other; p = 0.98, t-test, 2 sided

7. Secondary Outcome: Change in Hip Bone Mineral Density (BMD)
Description: BMD was measured using a Dual Energy X-ray Absorptiometry (DEXA) scan and reported by T-scores, measurements made of the hip bones using the scan. The T-score reflects how your bone density measurement compares to normal healthy adults. A normal bone density results in a T-score between +1.0 and -1.0. A T-score of less than or equal to -1.5 was used for this study to define the presence of osteopenia/osteoporosis. Osteopenia is a condition of decreased bone mass or density but not thin enough to be diagnosed as osteoporosis. Osteoporosis is a condition where bone mass/density has diminished to a level causing higher risk of fracture. The average change in T-score from baseline to one year is reported.
Time Frame: Baseline, 1 year post kidney transplant
Population: Per-protocol analysis. Not all subjects were able to undergo the DEXA scan of the hip at baseline and one-year [Control n = 41/Treatment n = 40].
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Immunosuppression Without Paricalcitol (Control) | Immunosuppression With Paricalcitol
Number analyzed (Participants) | 41 | 40
T-score | 0.15 (0.27) | 0.21 (0.36)
Statistical Analysis 1: Comparison: Immunosuppression Without Paricalcitol (Control) vs Immunosuppression With Paricalcitol; Test type: Superiority or Other; p = 0.41, t-test, 2 sided

8. Secondary Outcome: Number of Subjects Who Died or Lost Their Renal Graft During First Year
Description: The number of subject who died (or experienced failure of their kidney surgical graft) during the first year following kidney transplant are reported here.
Time Frame: Baseline to 1 year post kidney transplant
Population: Per-protocol analysis.
Measure: Number; unit: participants
Arm/Group | Immunosuppression Without Paricalcitol (Control) | Immunosuppression With Paricalcitol
Number analyzed (Participants) | 44 | 43
participants | 0 | 1

9. Secondary Outcome: Episodes of Acute Cellular Rejection (ACR) of the Renal Transplant
Description: The number of episodes of ACR, as proven by renal biopsy, were recorded.
Time Frame: Baseline to 1 year post kidney transplant
Population: Per-protocol analysis.
Measure: Number; unit: episodes
Arm/Group | Immunosuppression Without Paricalcitol (Control) | Immunosuppression With Paricalcitol
Number analyzed (Participants) | 44 | 43
episodes | 5 | 4

10. Secondary Outcome: Mean Estimated Glomerular Filtration Rate (eGFR) at One Year
Description: Glomerular filtration rate describes the amount that fluid is filtered through the kidney and can be estimated by using serum creatinine. eGFR is reported in milliliters per minute per 1.73 m^2 of body-surface area.
Time Frame: 1 year post kidney transplant
Population: Per-protocol analysis
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Immunosuppression Without Paricalcitol (Control) | Immunosuppression With Paricalcitol
Number analyzed (Participants) | 44 | 43
mL/min/1.73m^2 | 52.7 (14.1) | 51.2 (15.4)
Statistical Analysis 1: Comparison: Immunosuppression Without Paricalcitol (Control) vs Immunosuppression With Paricalcitol; Test type: Superiority or Other; p = 0.66, t-test, 2 sided

11. Secondary Outcome: Mean Change in Estimated Glomerular Filtration Rate (eGFR) Between 3 Weeks and 1 Year Post Transplant
Time Frame: 3 weeks, 1 year post kidney transplant
Population: Per-protocol analysis
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Immunosuppression Without Paricalcitol (Control) | Immunosuppression With Paricalcitol
Number analyzed (Participants) | 44 | 43
mL/min/1.73 m^2 | 7.4 (15.1) | 6.2 (10.4)
Statistical Analysis 1: Comparison: Immunosuppression Without Paricalcitol (Control) vs Immunosuppression With Paricalcitol; Test type: Superiority or Other; p = 0.66, t-test, 2 sided

12. Secondary Outcome: 24-hour Total Protein in the Urine at 1 Year Post Transplant
Description: A urine total protein test is conducted to detect excess protein in the urine. This test helps determine an individual's kidney functioning. Protein is not usually present in urine; therefore, presence of protein in the urine is a sign of abnormality. The quantity of protein in a sample of urine collected over 24-hour was measured and reported in milligrams per day.
Time Frame: 1 year post kidney transplant
Population: Per-protocol analysis. The 24-hour urine collection was not completed for all subjects.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Immunosuppression Without Paricalcitol (Control) | Immunosuppression With Paricalcitol
Number analyzed (Participants) | 40 | 36
mg/day | 420.8 (1052.3) | 159.4 (235.8)
Statistical Analysis 1: Comparison: Immunosuppression Without Paricalcitol (Control) vs Immunosuppression With Paricalcitol; Test type: Superiority or Other; p = 0.11, t-test, 2 sided

13. Secondary Outcome: Degree of Interstitial Fibrosis on Graft Biopsy at One Year
Description: Interstitial fibrosis refers to degree of scarring or fibrous tissue formed in the kidney. Renal pathologists reviewed biopsies of the subject's kidney grafts for fibrosis, with results expressed using the Banff schema; Quantitative criteria: ci0 = fibrosis observed in up to 5% of cortical area, ci1 = fibrosis in 6%-25% of cortical area (mild) , ci2 = fibrosis in 26%-50% of cortical area (moderate), ci3 = fibrosis in greater than 50% of cortical area (severe). The degree of interstital fibrosis for this study was defined and reported as follows: a Banff ci score of greater than 0 and less than 2 considered "mild" fibrosis and a ci score greater than or equal to 2 as "moderate to severe" fibrosis.
Time Frame: 1 year post kidney transplant
Population: Per-protocol analysis; graft biopsies were not available for all subjects
Measure: Number; unit: Participants
Arm/Group | Immunosuppression Without Paricalcitol (Control) | Immunosuppression With Paricalcitol
Number analyzed (Participants) | 38 | 38
Participants
  Mild fibrosis at 1 year | 19 (50) | 19 (50)
  Moderate to severe fibrosis at 1 year | 4 (10.5) | 0 (0)
Statistical Analysis 1: Comparison: Immunosuppression Without Paricalcitol (Control) vs Immunosuppression With Paricalcitol; The number of subjects with mild interstitial fibrosis (Banff ci score > 0 and < 2) at one year was compared between treatment groups; Test type: Superiority or Other; p = 1.0, t-test, 2 sided
Statistical Analysis 2: Comparison: Immunosuppression Without Paricalcitol (Control) vs Immunosuppression With Paricalcitol; The number of subjects with moderate to mild interstitial fibrosis (Banff ci score greater than or equal to 2) at one year was compared between treatment groups; Test type: Superiority or Other; p = 0.04, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and collected from baseline to 52 weeks post kidney transplant.
Description: Adverse events were determined based on changes in clinical symptoms and changes in laboratory results at various timepoints and during study visits. Mayo Clinic management programs currently in place for renal transplant recipients with specific laboratory abnormalities were used to diagnose and manage conditions.
Arm/Group | Immunosuppression Without Paricalcitol (Control) | Immunosuppression With Paricalcitol
Serious Adverse Events (participants affected / at risk) | 16/49 | 27/51
Other Adverse Events (participants affected / at risk) | 14/49 | 32/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunosuppression Without Paricalcitol (Control) (N=49) | Immunosuppression With Paricalcitol (N=51)
neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Orthostasis (Cardiac disorders) | 0 (0) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
fever (General disorders) | 1 (1) | 1 (1)
headache (General disorders) | 0 (0) | 1 (1)
malaise (General disorders) | 0 (0) | 1 (1)
liver cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
allergy to intravenous immunoglobulin (Immune system disorders) | 1 (1) | 0 (0)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
bone fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
right leg radicular pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
incidental renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
seizure (Nervous system disorders) | 0 (0) | 1 (1)
depression (Psychiatric disorders) | 1 (1) | 0 (0)
paranoia (Psychiatric disorders) | 0 (0) | 1 (1)
acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
hydronephrosis (Renal and urinary disorders) | 1 (1) | 4 (4)
bilateral native nephrectomy (Surgical and medical procedures) | 1 (1) | 4 (4)
hernia repair (Surgical and medical procedures) | 0 (0) | 4 (4)
hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
motor vehicle accident (Surgical and medical procedures) | 0 (0) | 1 (1)
ureteral revision (Surgical and medical procedures) | 0 (0) | 2 (2)
biopsy complication (Surgical and medical procedures) | 1 (1) | 0 (0)
pulmonary embolus (Vascular disorders) | 0 (0) | 2 (2)
peripheral vascular disease (Vascular disorders) | 0 (0) | 2 (2)
chylous ascitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
vertebral artery dissection (Vascular disorders) | 0 (0) | 1 (1)
hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
lymphocele (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
surgical incision pain (Surgical and medical procedures) | 1 (1) | 0 (0)
ureteric revision (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
wound complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus (Infections and infestations) | 1 (1) | 1 (1)
gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 1 (1) | 0 (0)
scrotal cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Turberculosis, Active (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0)
wound infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 5 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Immunosuppression Without Paricalcitol (Control) (N=49) | Immunosuppression With Paricalcitol (N=51)
Post transplant diabetes mellitus (Endocrine disorders) | 2 (2) | 4 (4)
diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
allergy to Bactrim (Immune system disorders) | 0 (0) | 1 (1)
gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
symptomatic hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fall in bathroom (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Re-operation (Surgical and medical procedures) | 0 (0) | 1/46 (1)
viral (BK) nephropathy (Infections and infestations) | 0 (0) | 1 (1)
BK viremia (Infections and infestations) | 4 (4) | 0 (0)
pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 1 (1) | 1 (1)
sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus viremia (Infections and infestations) | 0 (0) | 2 (2)
Clostridium difficile (Infections and infestations) | 0 (0) | 1 (1)
bladder urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
glomerulonephritis (Renal and urinary disorders) | 1 (1) | 1 (1)
Surgical Incision Pain (Surgical and medical procedures) | 1 (1) | 0 (0)
Urinary Tract Infections (Infections and infestations) | 0 (0) | 10 (11)
Wound Complication (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less